CLINICAL TRIAL: NCT07322172
Title: Pilot Study of Patient Navigation Intervention to Improve Follow-up Care for Patients With Urinary Stone Disease
Brief Title: Pilot Study of Patient Navigation for Kidney Stone Patients After ED Visits
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-45298; 1K23DK141906-01A1 (NIH)
Record Dates: First submitted 2026-01-02; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Navigation Intervention (Experimental)
  Interventions: Other: Patient Navigation

INTERVENTIONS:
Other: Patient Navigation — The intervention consists of a patient navigation program delivered by a patient navigator over approximately 12 weeks. Participants identified as high risk for loss to follow-up after an emergency department visit for kidney stone disease will receive individualized navigation support focused on identifying and addressing barriers to urology follow-up. Navigation activities may include care coordination support, appointment scheduling guidance, health education, linkage to existing institutional or community resources (transportation assistance or insurance enrollment support), and motivational support. The patient navigator will maintain regular contact with participants through in-person, phone, or virtual encounters, and navigation activities will be documented in a secure research database. The intervention is designed to support access to recommended care and does not alter clinical treatment decisions.

SUMMARY:
Patients who visit the emergency department for kidney stones are sometimes referred to urology for follow-up care but never complete that visit. Missing follow-up appointments can lead to worse outcomes, including recurrent pain, infection, or surgery. Research shows that patients who are socially or economically at risk (such as those with public insurance, lower income, or limited English proficiency) are more likely to experience these care gaps.

This study will pilot a patient navigation program designed to help patients with urinary stone disease (USD) attend their scheduled urology appointments after being seen in the Emergency Department. Using an electronic health record (EHR) based prediction model developed in earlier research, patients at higher risk for being lost to follow-up will be identified and invited to participate. Each participant will be paired with a trained patient navigator who will assess barriers to care, provide support, and maintain contact for about 12 weeks.

The goal of this study is to evaluate the outcomes and feasibility of this navigation intervention. Findings will help determine whether a larger study should test if this approach improves access to care and health outcomes for patients with kidney stones.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presentation to the Emergency Department with urinary stone disease
* Placement of an outpatient urology referral from the Emergency Department
* Identified as high risk for loss to follow-up based on the study's screening process

Exclusion Criteria:

* Age < 18 years
* Unable to provide informed consent
* Non-English-speaking
* No outpatient urology referral placed from the Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Completion of an outpatient urology follow-up visit within 12 weeks of emergency department discharge, assessed through review of the electronic health record. | From enrollment to the end of intervention at 12 weeks

SECONDARY OUTCOMES:
Acceptability of the Patient Navigation Intervention Measured by the Patient Navigation Process and Outcomes Measure (PNPOM) | From enrollment to the end of treatment at 12 weeks
  Acceptability will be assessed using the Patient Navigation Process and Outcomes Measure (PNPOM), a validated questionnaire administered to patient participants at the completion of the intervention. The PNPOM evaluates participants' perceptions of the navigation experience, including satisfaction, perceived usefulness, and support received. Responses are scored on a Likert-type scale, with higher scores indicating greater acceptability of the navigation intervention. The total score will be summarized descriptively to assess overall intervention acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: David Bayne, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Srirangapatanam S, Suarez P, Chi T, Neuhaus J, Stoller M, Scales S, Bayne D. EMR data enhances prediction accuracy for care delays compared to standard demographic data. Presented at: AUA 2024, San Antonio, Texas, May 3-6. Abstract MP40-08
- [Background] Suarez PA, Srirangapatanam S, Leng L, Momodu MM, Neuhaus J, Bayne DB. Enhancing surgical efficiency: predicting same-day cancellations in urologic procedures. World J Urol. 2025 Dec 17;44(1):48. doi: 10.1007/s00345-025-06155-6. PMID 41405624